CLINICAL TRIAL: NCT07123467
Title: Cannabidiol-Enhanced Cognitive Behavioral Therapy for Generalized Anxiety Disorder
Brief Title: Cannabidiol-Assisted Learning for Managing Generalized Anxiety Disorder
Acronym: CALM
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Hilary Marusak, Associate Professor, Department of Psychiatry and Behavioral Neuroscience, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-24-11-7333; R61MH137105 (NIH)
Record Dates: First submitted 2025-08-02; First posted 2025-08-14 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-08

CONDITIONS: Generalized Anxiety Disorder (GAD); Anxiety Disorders
Keywords: Cannabidiol; EPIDIOLEX; Cognitive Behavioral Therapy; Generalized Anxiety Disorder; functional magnetic resonance imaging
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants, therapists, study staff, and outcomes assessors will be blinded to treatment assignment. Only the principal investigators hold the randomization and blinding key. Placebo is a matched oral solution designed to mimic EPIDIOLEX® in appearance, taste, and smell to maintain effective blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Brief Cognitive Behavioral Therapy + Moderate-Dose Cannabidiol (Experimental): Participants will receive a 5-week course of brief cognitive behavioral therapy (CBT) combined with oral cannabidiol (EPIDIOLEX®) at a moderate dose. Dosing starts at 5 milligram/kilogram/day and titrates to 10 milligram/kilogram/day (divided twice a day) after 6 days. Cannabidiol is administered chronically throughout CBT to examine target engagement and symptom outcomes.
  Interventions: Drug: Moderate-Dose Cannabidiol
- Brief Cognitive Behavioral Therapy + Low-Dose Cannabidiol (Experimental): Participants will receive a 5-week course of brief cognitive behavioral therapy (CBT) combined with a lower dose of oral cannabidiol (EPIDIOLEX®), maintained at 5 milligram/kilogram/day (divided twice a day) throughout the treatment period. No titration is required.
  Interventions: Drug: Low-Dose Cannabidiol
- Brief Cognitive Behavioral Therapy + Placebo Titrated to Match Moderate-Dose Cannabidiol (Placebo Comparator): Participants will receive a 5-week course of brief cognitive behavioral therapy (CBT) combined with a matched placebo oral solution. The placebo mimics the appearance, smell, and taste of EPIDIOLEX®. For blinding the moderate dose cannabidiol arm, dosing starts at 5 milligram/kilogram/day and titrates to 10 milligram/kilogram/day (divided twice a day) after 6 days.
  Interventions: Drug: Placebo Matched to Moderate-Dose Cannabidiol
- Brief Cognitive Behavioral Therapy + Placebo Titrated to Match Low-Dose Cannabidiol (Placebo Comparator): Participants will receive a 5-week course of brief cognitive behavioral therapy (CBT) combined with a matched placebo oral solution. The placebo mimics the appearance, smell, and taste of EPIDIOLEX®. For blinding the low-dose cannabidiol arm, dosing is maintained at 5 milligram/kilogram/day (divided twice a day) throughout the treatment period. No titration is required.
  Interventions: Drug: Placebo Matched to Low-Dose Cannabidiol

INTERVENTIONS:
Drug: Low-Dose Cannabidiol — Oral cannabidiol solution (EPIDIOLEX®) administered as an adjunct to cognitive behavioral therapy. Low-dose participants receive 5 milligram/kilogram/day throughout. The intervention targets emotion regulation circuitry and symptom improvement.
  Other Names: EPIDIOLEX®
  Arms: Brief Cognitive Behavioral Therapy + Low-Dose Cannabidiol
Drug: Placebo Matched to Moderate-Dose Cannabidiol — The placebo mimics the appearance, smell, and taste of EPIDIOLEX®. For blinding the moderate-dose cannabidiol arm, dosing starts at 5 mg/kg/day and titrates to 10 milligram/kilogram/day (divided twice a day) after 6 days.
  Arms: Brief Cognitive Behavioral Therapy + Placebo Titrated to Match Moderate-Dose Cannabidiol
Drug: Moderate-Dose Cannabidiol — Oral cannabidiol solution (EPIDIOLEX®) administered as an adjunct to cognitive behavioral therapy. Moderate-dose participants receive 5 milligram/kilogram/day for 6 days, then titrate to 10 milligram/kilogram/day. The intervention targets emotion regulation circuitry and symptom improvement.
  Other Names: EPIDIOLEX®
  Arms: Brief Cognitive Behavioral Therapy + Moderate-Dose Cannabidiol
Drug: Placebo Matched to Low-Dose Cannabidiol — The placebo mimics the appearance, smell, and taste of EPIDIOLEX®. For blinding the low-dose cannabidiol arm, dosing is maintained at 5 milligram/kilogram/day (divided twice a day) throughout the treatment period. No titration is required.
  Arms: Brief Cognitive Behavioral Therapy + Placebo Titrated to Match Low-Dose Cannabidiol

SUMMARY:
This randomized, double-blind, placebo-controlled clinical trial investigates the use of Food and Drug Administration (FDA)-approved cannabidiol (EPIDIOLEX®) as an adjunct to cognitive behavioral therapy (CBT) in adults with generalized anxiety disorder (GAD). The study aims to evaluate whether cannabidiol-assisted CBT enhances emotion regulation via dorsomedial prefrontal cortex (dmPFC) activation and improves anxiety symptom outcomes compared to CBT with placebo.

DETAILED DESCRIPTION:
The study is a randomized, double-blind, placebo-controlled clinical trial evaluating cannabidiol (CBD) as an adjunct to cognitive behavioral therapy (CBT) for treating generalized anxiety disorder (GAD) in adults aged 18-45. Participants will be randomly assigned to one of four arms: (1) Brief CBT with moderate-dose EPIDIOLEX® (10 milligrams(mg)/kilograms(kg)/day), (2) Brief CBT with low-dose EPIDIOLEX® (5 mg/kg/day), (3) Brief CBT with matched placebo with dosing matched to the moderate-dose EPIDIOLEX®, or 4) Brief CBT with matched placebo with dosing matched to the low-dose EPIDIOLEX®. The trial uses a neurobiologically informed experimental medicine approach to evaluate target engagement in the dorsomedial prefrontal cortex (dmPFC) during an emotion regulation functional magnetic resonance imaging (fMRI) task before and after treatment. Primary outcomes include change in dmPFC activation, while secondary outcomes include anxiety symptom severity, treatment tolerability, and plasma concentrations of cannabidiol and related biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed
* Age 18-45 years at enrollment
* Able to consent to the study
* Agree to adhere to lifestyle considerations throughout study duration
* Generally medically and neurologically healthy, including no evidence of intellectual disability or serious cognitive impairment
* Have a current generalized anxiety disorder (GAD) diagnosis according to the The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria and/or total scores ≥ 8 on the 7-Item Generalized Anxiety Disorders Scale (GAD-7)

Exclusion Criteria:

* Clinically significant medical or neurologic condition or neurocognitive dysfunction that would affect function and/or task performance and/or interfere with the study protocol
* Any current (or within past 2 months) medical condition requiring medication that would interact with cannabidiol or interfere with the study protocol
* Risk of harm to self or others that requires immediate intervention
* Presence of contraindications, current or past allergic or adverse reaction, or known sensitivity to cannabinoid-like substances or components of EPIDIOLEX®
* Positive drug screen or alcohol breathalyzer
* Unwilling/unable to sign informed consent document
* Currently pregnant (positive pregnancy test), planning pregnancy, or lactating (women),
* Under 18 or over 45 years of age
* Traumatic brain injury, as defined by The American Congress of Rehabilitation as a person who has had a traumatically induced physiological disruption of brain function (i.e., the head being struck, the head striking an object, and/or the brain undergoing an acceleration/deceleration movement [i.e., whiplash] without direct external trauma to the head), as manifested by at least one of the following: any loss of consciousness; any loss of memory for events immediately before or after the injury; any alteration in mental status at the time of the incident; or focal neurological deficits that may or may not be transient)
* Inability to tolerate small, enclosed spaces without anxiety (e.g. claustrophobia), as determined by self-report and/or a preliminary session in a mock scanner
* Presence of ferrous-containing metals within the body (e.g., aneurysm clips, shrapnel/retained particles)
* Receiving concurrent psychotherapy or have received psychotherapy, including for research purposes, within the past year
* Current moderate or severe alcohol/drug use disorder or in the past 8 weeks
* Current or past diagnosis of bipolar and other related disorders, schizophrenia spectrum, or other psychotic disorders;
* GAD-7 score < 8
* Use of medications known to have severe drug interactions with cannabidiol or that are strong inducers of cytochrome P450 3A4 (CYP3A4) or cytochrome P450 2C19 (CYP2C19)
* Visual impairment
* Baseline labs 3 times outside of normal range
* Use of as needed anti-anxiety medications (e.g., benzodiazepines), unstable dose of other psychoactive drug (i.e., < 4 weeks), or intention to start new treatment during this trial
* Current or past-month use of cannabis, or a tetrahydrocannabinol (THC) or cannabidiol-containing product (self-report and urine drug screen)
* Current or past-month coronavirus disease 2019 (COVID-19) diagnosis or febrile illness
* Treatment with another investigational drug or intervention within the past month
* Difficulty with or inability to comply with the complete clinical trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in dorsomedial prefrontal cortex activation when reappraising negative images | Baseline to post-treatment (~Week 5)
  Within-participant change in dorsomedial prefrontal cortex (dmPFC) activation will be calculated as post-treatment minus baseline values during an explicit emotion regulation task (Reappraise > Maintain contrast). Measured using blood-oxygen-level-dependent (BOLD) signal from multi-echo functional magnetic resonance imaging (fMRI).

SECONDARY OUTCOMES:
Post-treatment dorsomedial prefrontal cortex activation when reappraising negative images | Post-treatment (~Week 5)
  Post-treatment dorsomedial prefrontal cortex (dmPFC) activation during an explicit emotion regulation task (Reappraise > Maintain contrast). Measured using blood-oxygen-level-dependent (BOLD) signal from multi-echo functional magnetic resonance imaging (fMRI).
Post-treatment amygdala activation when reappraising negative images | Post-treatment (~Week 5)
  Post-treatment amygdala activation during an explicit emotion regulation task (Reappraise > Maintain contrast). Measured using blood-oxygen-level-dependent (BOLD) signal from multi-echo functional magnetic resonance imaging (fMRI).
Change in amygdala activation when reappraising negative images | Baseline to post-treatment (~Week 5)
  Within-participant change in amygdala activation will be calculated as post-treatment minus baseline values during an explicit emotion regulation task (Reappraise > Maintain contrast). Measured using blood-oxygen-level-dependent (BOLD) signal from multi-echo functional magnetic resonance imaging (fMRI).
Post-treatment hippocampal activation when reappraising negative images | Post-treatment (~Week 5)
  Post-treatment hippocampal activation during an explicit emotion regulation task (Reappraise > Maintain contrast). Measured using blood-oxygen-level-dependent (BOLD) signal from multi-echo functional magnetic resonance imaging (fMRI).
Change in hippocampal activation when reappraising negative images | Baseline to post-treatment (~Week 5)
  Within-participant change in hippocampal activation will be calculated as post-treatment minus baseline values during an explicit emotion regulation task (Reappraise > Maintain contrast). Measured using blood-oxygen-level-dependent (BOLD) signal from multi-echo functional magnetic resonance imaging (fMRI).
Post-treatment inferior frontal gyrus activation when reappraising negative stimuli | Post-treatment (~Week 5)
  Post-treatment inferior frontal gyrus activation during an explicit emotion regulation task (Reappraise > Maintain contrast). Measured using blood-oxygen-level-dependent (BOLD) signal from multi-echo functional magnetic resonance imaging (fMRI).
Change in inferior frontal gyrus activation when reappraising negative images | Baseline to post-treatment (~Week 5)
  Within-participant change in inferior frontal gyrus activation will be calculated as post-treatment minus baseline values during an explicit emotion regulation task (Reappraise > Maintain contrast). Measured using blood-oxygen-level-dependent (BOLD) signal from multi-echo functional magnetic resonance imaging (fMRI).
Post-treatment anterior insula activation when reappraising negatives images | Post-treatment (~Week 5)
  Post-treatment anterior insula activation during an explicit emotion regulation task (Reappraise > Maintain contrast). Measured using blood-oxygen-level-dependent (BOLD) signal from multi-echo functional magnetic resonance imaging (fMRI).
Change in anterior insula activation when reappraising negative images | Baseline to post-treatment (~Week 5)
  Within-participant change in anterior insula activation will be calculated as post-treatment minus baseline values during an explicit emotion regulation task (Reappraise > Maintain contrast). Measured using blood-oxygen-level-dependent (BOLD) signal from multi-echo functional magnetic resonance imaging (fMRI).
Change in plasma concentration of anandamide from baseline to post-treatment | Baseline and post-treatment (~Week 5)
  Plasma anandamide levels will be measured via liquid chromatography-tandem mass spectrometry (LC-MS/MS) at baseline and post-treatment. Change will be calculated as post-treatment minus baseline values (nanogram per milliliter).
Change in plasma concentration of 2-arachidonoylglycerol (2-AG) from baseline to post-treatment | Baseline and post-treatment (~Week 5)
  Plasma 2-arachidonoylglycerol (2-AG) levels will be measured via liquid chromatography-tandem mass spectrometry (LC-MS/MS) at baseline and post-treatment. Change will be calculated as post-treatment minus baseline values (nanogram per milliliter).
Change in plasma concentration of cannabidiol from baseline to post-treatment | Baseline and post-treatment (~Week 5)
  Plasma cannabidiol levels will be measured via liquid chromatography-tandem mass spectrometry (LC-MS/MS) at baseline and post-treatment. Change will be calculated as post-treatment minus baseline values (nanogram per milliliter).
Change in plasma concentration of 7-hydroxy-cannabidiol (7-OH-CBD) from baseline to post-treatment | Baseline and post-treatment (~Week 5)
  7-hydroxy-cannabidiol (7-OH-CBD; active metabolite) levels will be measured via liquid chromatography-tandem mass spectrometry (LC-MS/MS) at baseline and post-treatment. Change will be calculated as post-treatment minus baseline values (nanogram per milliliter).
Post-treatment dorsomedial prefrontal cortex activation during implicit emotion regulation | Post-treatment (~Week 5)
  Post-treatment dorsomedial prefrontal cortex (dmPFC) activation during an implicit emotion regulation task. Measured using blood-oxygen-level-dependent (BOLD) signal from multi-echo functional magnetic resonance imaging (fMRI).
Change in dorsomedial prefrontal cortex activation during implicit emotion regulation | Baseline to post-treatment (~Week 5)
  Within-participant change in dorsomedial prefrontal cortex (dmPFC) activation will be calculated as post-treatment minus baseline values during an implicit emotion regulation task. Measured using blood-oxygen-level-dependent (BOLD) signal from multi-echo functional magnetic resonance imaging (fMRI).
Post-treatment ventromedial prefrontal cortex activation during implicit emotion regulation | Post-treatment (~Week 5)
  Post-treatment ventromedial prefrontal cortex (vmPFC) activation during implicit emotion regulation. Measured using blood-oxygen-level-dependent (BOLD) signal from multi-echo functional magnetic resonance imaging (fMRI).
Change in ventromedial prefrontal cortex activation during implicit emotion regulation | Baseline to post-treatment (~Week 5)
  Within-participant change in ventromedial prefrontal cortex (vmPFC) activation will be calculated as post-treatment minus baseline values during an implicit emotion regulation task. Measured using blood-oxygen-level-dependent (BOLD) signal from multi-echo functional magnetic resonance imaging (fMRI).
Change in depressive symptom severity | Baseline and post-treatment (~Week 5)
  Change in depressive symptom severity will be assessed using the 9-item Patient Health Questionnaire (PHQ-9), a validated self-report instrument that measures symptoms of depression over the past two weeks. Each item is rated on a 0-3 scale, producing a total score ranging from 0 to 27, with higher scores indicating greater severity. Scores will be collected at baseline and post-treatment. Change will be calculated as post-treatment minus baseline score.

CONTACTS AND LOCATIONS:
Overall Officials: Hilary Marusak, PhD, Principal Investigator — Wayne State University; Christine Rabinak, PhD, MBA, Principal Investigator — Wayne State Universty; Leslie Lundahl, PhD, Principal Investigator — Wayne State University
Locations (2):
- United States (2):
  - Wayne State University Eugene Applebaum College of Pharmacy & Health Sciences, Detroit, Michigan
  - Wayne State University School of Medicine, Tolan Park Medical Building, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) supporting the primary and secondary outcomes - including symptom measures, functional magnetic resonance imaging activation and connectivity metrics, and plasma concentrations of cannabidiol and metabolites - will be shared.
Time Frame: Individual participant data (IPD) will be shared beginning 12 months after publication of the primary study results and will remain available for at least 5 years thereafter.
Access Criteria: Data will be made available to qualified researchers via the National Institute of Mental Health Data Archive (NDA). Access will be granted to investigators with an approved research proposal and appropriate data use agreement.
URL: https://nda.nih.gov

REFERENCES:
- [Background] Zabik NL, Iadipaolo A, Peters CA, Baglot SL, Hill MN, Rabinak CA. Dose-dependent effect of acute THC on extinction memory recall and fear renewal: a randomized, double-blind, placebo-controlled study. Psychopharmacology (Berl). 2024 Oct 16:10.1007/s00213-024-06702-w. doi: 10.1007/s00213-024-06702-w. Online ahead of print. PMID 39412674
- [Background] Zabik NL, Rabinak CA, Peters CA, Iadipaolo A. Cannabinoid modulation of corticolimbic activation during extinction learning and fear renewal in adults with posttraumatic stress disorder. Neurobiol Learn Mem. 2023 May;201:107758. doi: 10.1016/j.nlm.2023.107758. Epub 2023 Apr 22. PMID 37088409
- [Background] Pacitto R, Peters C, Iadipaolo A, Rabinak CA. Cannabinoid modulation of brain activation during volitional regulation of negative affect in trauma-exposed adults. Neuropharmacology. 2022 Nov 1;218:109222. doi: 10.1016/j.neuropharm.2022.109222. Epub 2022 Aug 15. PMID 35981598
- [Background] Mayo LM, Rabinak CA, Hill MN, Heilig M. Targeting the Endocannabinoid System in the Treatment of Posttraumatic Stress Disorder: A Promising Case of Preclinical-Clinical Translation? Biol Psychiatry. 2022 Feb 1;91(3):262-272. doi: 10.1016/j.biopsych.2021.07.019. Epub 2021 Jul 24. PMID 34598785
- [Background] Gorka SM, Phan KL, Lyons M, Mori S, Angstadt M, Rabinak CA. Cannabinoid Modulation of Frontolimbic Activation and Connectivity During Volitional Regulation of Negative Affect. Neuropsychopharmacology. 2016 Jun;41(7):1888-96. doi: 10.1038/npp.2015.359. Epub 2015 Dec 9. PMID 26647971
- [Background] Gowatch LC, Evanski JM, Ely SL, Zundel CG, Bhogal A, Carpenter C, Shampine MM, O'Mara E, Mazurka R, Barcelona J, Mayo LM, Marusak HA. Endocannabinoids and Stress-Related Neurospsychiatric Disorders: A Systematic Review and Meta-Analysis of Basal Concentrations and Response to Acute Psychosocial Stress. Cannabis Cannabinoid Res. 2024 Oct;9(5):1217-1234. doi: 10.1089/can.2023.0246. Epub 2024 Apr 29. PMID 38683635